CLINICAL TRIAL: NCT05568784
Title: Quadriceps Activation Comparative Analysis Based on Positioning of the Ankle During Supine Straight Leg Raise and Quad Set
Brief Title: Straight Leg Raise Continuation
Acronym: SLR
Status: Recruiting | Type: Observational
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Florida (Other)
Responsible Party: Sponsor
Other Study IDs: SLR Continuation
Record Dates: First submitted 2022-09-30; First posted 2022-10-06 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Quadriceps Muscle Atrophy; Leg Injury
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Participants: Patients without pre-existing lower extremity injury that may inhibit response to testing
  Interventions: Other: Straight Leg Raise exercise
- Participants with Knee Arthroscopy: Patients who have recently suffered knee injury that required arthroscopic surgery
  Interventions: Other: Straight Leg Raise exercise

INTERVENTIONS:
Other: Straight Leg Raise exercise — Patient lying supine will lift leg to the height of the contralateral knee flexed to 90 degrees with the ankle positioned and tested in all three positions (dorsiflexion, neutral, and plantarflexion)

SUMMARY:
The goal of this study is to compare quadriceps muscle activation in patients recovering from lower extremity injury, such as an ACL tear. Specifically, the main objectives are as follows:

* Determine the effects of ankle positioning on quad muscle activation during straight leg raise exercises performed while the patient is lying on his or her back
* Determine if there is a difference between ankle positioning on quad muscle activation during straight leg raise exercises performed while the patient is lying on his or her back, comparing healthy versus post-operative participants

DETAILED DESCRIPTION:
Returning quadriceps neuromuscular control and preventing atrophy is an area of intense current interest in orthopedic rehabilitation and recovery science. It is clear that returning full autonomous control of the quadriceps, including the vastus medialis obliqus (VMO), at full knee extension is an important factor in rehab and dysfunction of the quadriceps leads to a loss of physical performance and self-reported function. Quadriceps function is critical for optimal ambulation patterns and eccentric control is essential for the weight acceptance phase of gait.

Quadriceps atrophy is one of the most common post-operative side effects of anterior cruciate ligament (ACL) reconstruction, total knee arthroplasty, and many other surgeries including meniscal repairs, patella realignment procedures, and microfracture procedures. Due to the swelling within the joint after injury or surgery to the knee, the joint inflammation cascade occurs and leads to the quadriceps being arthrogenically inhibited by spinal neuron inhibition as a protective mechanism. These neural changes usually lead to decreased voluntary quadriceps contraction. Additional contributions of inhibition from post-operative pain, patient apprehension, and surgical procedure requiring protection of the repaired tissue. The sooner one regains control of the quadriceps muscles the less atrophy occurs, reductions in strength are minimized, and the more optimal the outcome is achieved for patient recovery.

Studies have shown that neuromuscular electrical stimulation (NMES), Transcutaneous electrical nerve stimulation (TENS), and biofeedback techniques can limit post-operative quadriceps atrophy and can return strength of the quadriceps back to normative values faster than without those techniques and traditional therapeutic exercise and have better long-term outcomes based on pain, functional outcomes, and return to sport participation rates.

Irradiation effect is a proprioceptive neuromuscular facilitation technique that causes an overflow of neuronal energy from distal to proximal muscles to increase muscle activity of a targeted muscle. This technique can be used to selectively recruit weaker motor units through the application of resistance or stimulation. By inducing a stronger contractile force of the quadriceps, our hope is to return quadriceps function to normal quicker with less atrophy and greater strength.

The investigators hypothesize that ankle positioning in maximal dorsiflexion (DF) changes the quantity of contraction as a percent of the reference voluntary contraction when performing a supine straight leg raise compared with having the foot in neutral (0°), relaxed, and plantarflexed (PF) positions. This may help provide insight into proper instruction and cuing for patients to return quadriceps neuromuscular control sooner and thus limiting quadriceps atrophy.

ELIGIBILITY:
(All Participants)

Inclusion Criteria:

* Males and females ages 18-55

Exclusion Criteria:

* History of diagnosed cancer, neurological disorder, peripheral nerve injury affecting the lower limb or injury to the lower spine with radicular symptoms, which may affect quadriceps activation
* History of musculoskeletal injury to the quadriceps that may affect ability to maintain muscle contractions without excessive fatigue or discomfort

(Healthy Participants)

Exclusion Criteria:

* Injury to the knee or quadriceps muscle group within the past 12 months to the tested side
* History of lower extremity orthopedic surgery in the past 12 months to the tested side

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of two groups of 50 individual participants each. These groups are healthy participants and participants who have recently undergone knee arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-11 (Actual); Primary Completion 2024-04-03 (Estimated); Study Completion 2024-07-03 (Estimated)

PRIMARY OUTCOMES:
Noraxon Ultium EMG | Within first 28 days post-op (Arthroscopy patients); healthy patients tested at enrollment
  Visually monitors and records electromagnetic signals from muscle activation using diodes placed on patient

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Opitz, PT, DPT, Principal Investigator — Physical Therapist
Locations (1):
- Andrews Research and Education Foundation, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harkey MS, Gribble PA, Pietrosimone BG. Disinhibitory interventions and voluntary quadriceps activation: a systematic review. J Athl Train. 2014 May-Jun;49(3):411-21. doi: 10.4085/1062-6050-49.1.04. Epub 2014 Feb 3. PMID 24490843
- [Background] Lewek MD, Rudolph KS, Snyder-Mackler L. Quadriceps femoris muscle weakness and activation failure in patients with symptomatic knee osteoarthritis. J Orthop Res. 2004 Jan;22(1):110-5. doi: 10.1016/S0736-0266(03)00154-2. PMID 14656668
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Background] Suter E, Herzog W, Bray RC. Quadriceps inhibition following arthroscopy in patients with anterior knee pain. Clin Biomech (Bristol). 1998 Jun;13(4-5):314-319. doi: 10.1016/s0268-0033(98)00098-9. PMID 11415802
- [Background] Palmieri RM, Tom JA, Edwards JE, Weltman A, Saliba EN, Mistry DJ, Ingersoll CD. Arthrogenic muscle response induced by an experimental knee joint effusion is mediated by pre- and post-synaptic spinal mechanisms. J Electromyogr Kinesiol. 2004 Dec;14(6):631-40. doi: 10.1016/j.jelekin.2004.06.002. PMID 15491837
- [Background] Hart JM, Pietrosimone B, Hertel J, Ingersoll CD. Quadriceps activation following knee injuries: a systematic review. J Athl Train. 2010 Jan-Feb;45(1):87-97. doi: 10.4085/1062-6050-45.1.87. PMID 20064053
- [Background] Hopkins J, Ingersoll CD. Arthrogenic muscle inhibition: A limiting factor in joint rehabilitation. Journal of Sport Rehabilitation. 2000;9(2):135-159.
- [Background] Palmieri RM, Weltman A, Edwards JE, Tom JA, Saliba EN, Mistry DJ, Ingersoll CD. Pre-synaptic modulation of quadriceps arthrogenic muscle inhibition. Knee Surg Sports Traumatol Arthrosc. 2005 Jul;13(5):370-6. doi: 10.1007/s00167-004-0547-z. Epub 2005 Feb 1. PMID 15685462
- [Background] Pietrosimone BG, Grindstaff TL, Linens SW, Uczekaj E, Hertel J. A systematic review of prophylactic braces in the prevention of knee ligament injuries in collegiate football players. J Athl Train. 2008 Jul-Aug;43(4):409-15. doi: 10.4085/1062-6050-43.4.409. PMID 18668174
- [Background] Palmieri-Smith RM, Kreinbrink J, Ashton-Miller JA, Wojtys EM. Quadriceps inhibition induced by an experimental knee joint effusion affects knee joint mechanics during a single-legged drop landing. Am J Sports Med. 2007 Aug;35(8):1269-75. doi: 10.1177/0363546506296417. Epub 2007 Jan 23. PMID 17244901
- [Background] Torry MR, Decker MJ, Viola RW, O'Connor DD, Steadman JR. Intra-articular knee joint effusion induces quadriceps avoidance gait patterns. Clin Biomech (Bristol). 2000 Mar;15(3):147-59. doi: 10.1016/s0268-0033(99)00083-2. PMID 10656976
- [Background] Panariello RA, Stump TJ, Allen AA. Rehabilitation and Return to Play Following Anterior Cruciate Ligament Reconstruction. Operative Techniques in Sports Medicine. 2017;25(3):181-193.
- [Background] Hopf HC, Schlegel HJ, Lowitzsch K. Irradiation of voluntary activity to the contralateral side in movements of normal subjects and patients with central motor disturbances. Eur Neurol. 1974;12(3):142-7. doi: 10.1159/000114613. No abstract available. PMID 4426322
- [Background] Moore JC. Excitation overflow: an electromyographic investigation. Arch Phys Med Rehabil. 1975 Mar;56(3):115-20. PMID 1119917
- [Background] Shimura K, Kasai T. Effects of proprioceptive neuromuscular facilitation on the initiation of voluntary movement and motor evoked potentials in upper limb muscles. Hum Mov Sci. 2002 Apr;21(1):101-13. doi: 10.1016/s0167-9457(01)00057-4. PMID 11983436
- [Background] Choi SA, Cynn HS, Yoon TL, Choi WJ, Lee JH. Effects of Ankle Dorsiflexion on Vastus Medialis Oblique and Vastus Lateralis Muscle Activity During Straight Leg Raise Exercise with Hip External Rotation in Patellofemoral Pain Syndrome. Journal of Musculoskeletal Pain. 2014;22(3):260-267.
- [Background] Holm B, Kristensen MT, Bencke J, Husted H, Kehlet H, Bandholm T. Loss of knee-extension strength is related to knee swelling after total knee arthroplasty. Arch Phys Med Rehabil. 2010 Nov;91(11):1770-6. doi: 10.1016/j.apmr.2010.07.229. PMID 21044725
- [Background] Hurley MV, Jones DW, Newham DJ. Arthrogenic quadriceps inhibition and rehabilitation of patients with extensive traumatic knee injuries. Clin Sci (Lond). 1994 Mar;86(3):305-10. doi: 10.1042/cs0860305. PMID 8156741
- [Background] Pietrosimone BG, Saliba SA, Hart JM, Hertel J, Kerrigan DC, Ingersoll CD. Effects of transcutaneous electrical nerve stimulation and therapeutic exercise on quadriceps activation in people with tibiofemoral osteoarthritis. J Orthop Sports Phys Ther. 2011 Jan;41(1):4-12. doi: 10.2519/jospt.2011.3447. Epub 2010 Dec 31. PMID 21282869

DOCUMENTS (2):
  • Study Protocol (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT05568784/Prot_000.pdf
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT05568784/ICF_001.pdf